CLINICAL TRIAL: NCT06054035
Title: SGLT2 Inhibition in Addition to Lifestyle Intervention and Risk for Complications in Subtypes of Patients With Prediabetes - a Randomized, Placebo Controlled, Multi-center Trial
Brief Title: SGLT2 Inhibition in Addition to Lifestyle Intervention and Risk for Complications in Subtypes of Patients With Prediabetes
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); German Center for Diabetes Research (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LIFETIME
Record Dates: First submitted 2023-09-06; First posted 2023-09-26 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Type2diabetes; PreDiabetes; Renal Failure
MeSH Terms: conditions — Prediabetic State; Renal Insufficiency | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Randomization will be performed stratified by prediabetes cluster.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Forxiga®) and lifestyle counselling (Experimental)
  Interventions: Drug: Dapagliflozin (Forxiga®); Behavioral: Lifestyle Intervention
- Placebo matching Dapaglifolzin and lifestyle counselling (Placebo Comparator)
  Interventions: Drug: Placebo matching Dapaglifolzin; Behavioral: Lifestyle Intervention

INTERVENTIONS:
Drug: Dapagliflozin (Forxiga®) — Dapagliflozin 10 mg once daily for 6 months. Route of administration: oral.
  Arms: Dapagliflozin (Forxiga®) and lifestyle counselling
Drug: Placebo matching Dapaglifolzin — Placebo matching Dapaglifolzin once daily for 6 months. Route of administration: oral.
  Arms: Placebo matching Dapaglifolzin and lifestyle counselling
Behavioral: Lifestyle Intervention — Patients receive a conventional lifestyle intervention (one in depth individual session at the beginning and standard care information on a healthy lifestyle at every visit thereafter).

SUMMARY:
More than 50% of patients with type 2 diabetes develop micro- and/or macrovascular complications during the course of the disease. Additionally, many patients at risk for diabetes develop metabolically driven complications including kidney and heart disease. Thus, it is of utmost importance to improve prevention of T2D and with this complications. Remission of prediabetes, i.e. normalization of hyperglycemia by means of lifestyle intervention is one of the most effective ways to prevent the development of T2D and complications. Novel sub-phenotyping analysis identified clusters of risk for diabetes associated with different complications, opening opportunities to new therapeutic approaches, despite and in addition to lifestyle changes. So far, pharmacological therapy is not indicated for patients with prediabetes. Remission of hyperglycemia associated with prediabetes during lifestyle interventions not only prevents T2D but is also linked with reduced albuminuria and lower microvascular and kidney complications. Thus, reaching normoglycemia (i.e. prediabetes remission) is important for reducing the risk of (pre-)diabetes-associated complications including micro- and even macrovascular disease. In patients with T2D, recent data show that dapagliflozin can improve diabetes remission, and thus, likely complications. However, to date no data have assessed whether or not this is also true in patients with hyperglycemia related to prediabetes which, as outlined above, already causes different complications.

Subphenotyping of patients with newly onset diabetes suggests that for some individuals, it would be too late to start interventions against dagainst complications at the time of diagnosis of type 2 diabetes. Therefore, individuals at elevated risk to develop T2D and complications should receive preventive measures well before the diagnosis of T2D. This study will provide evidence whether such an early intervention contributes to the remission of hyperglycemia related to prediabetes to protect from associated complications such as renal disease. The studied population will comprise individuals who have hyperglycemia in the range of prediabetes and are thus prone to not only develop T2D, but also early nephropathy but in clinical practice do not receive medical treatment due to the early stage of the disease. These subjects will receive Dapagliflozin 10 mg or Placebo for 6 months. The placebo treatment arm reflects current practice. In order guarantee a benefit the patients in the placebo arm will receive a lifestyle intervention.

ELIGIBILITY:
Inclusion criteria:

1. Male, female or intersexualpatients aged between 35 and 75 years (including)
2. Prediabetes (defined by one of the following: FG ≥ 100 mg/dL or 2h OGTT glucose ≥ 140 mg/dL)
3. BMI ≥20 kg/m2
4. TSH within normal range
5. Ability to understand and follow study-related instructions
6. Negative pregnancy test for premenopausal women (blood)
7. Patients who are receiving thyroid replacement therapy must be on a stable treatment regimen for at least 3 months prior to the screening visit (V-1)
8. Patients who are receiving antihypertensive medication such as mineralocorticoid receptor antagonists must be on a stable treatment regimen for at least 6 weeks prior to the screening visit (V-1)
9. Patients who are treated antihypertensive medication such as ACE inhibitors and AT1receptor antagonists, thiazides as well as loop diuretics must be on stable treatment for at least 2 weeks
10. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures.
11. Patients will not be included in the study if, in the opinion of the investigator participation will lead to an unacceptable risk to the subjects' safety or well-being

Exclusion Criteria

1. Manifest diabetes mellitus
2. eGFR (as calculated by the CKD-EPI equation) < 60 ml/min/1.73 m2
3. all glucose altering medications (including current therapy with dapagliflozin or empagliflozin or any other SGLT2-Inhibitor)
4. Symptomatic chronic congestive heart disease
5. New diuretic or antihypertensive medication or dosing changes within the last 2 weeks, for aldosterone antagonists within the last 6 weeks
6. known or suspected orthostatic proteinuria
7. any acute severe or chronic severe illness, including the following: malignant disease ongoing or < 5 years ago, unstable cardiovascular disease or procedure within 3 months prior to enrolment or expected to require coronary revascularisation procedure
8. history of or current therapy for congestive heart failure (NYHA III and IV), pacemaker or aortic stenosis > II°
9. acute pancreatic disease (i.e. elevated lipase 3x ULN)
10. rapidly progressing renal disease or anuria
11. known HIV infection or positive HIV test at screening
12. history of or planned organ transplantation
13. history or presence of inflammatory bowel disease or other severe gastrointestinal diseases, particularly those which may impact gastric emptying, such as gastroparesis or pyloric stenosis
14. relevant hepatic disease, including, but not limited to, acute hepatitis, chronic active hepatitis, or severe hepatic insufficiency, including patients with alanine aminotransferase and/or aspartate aminotransferase > 3 x upper limit of normal and/or total bilirubin (TB) > 2 mg/dL (> 34.2 μmol/L) (patients with TB > 2 mg/dL [> 34.2 μmol/L] and documented Gilbert's syndrome will be allowed to participate).
15. treatment with glucocorticoids
16. antibiotic treatment within the last 4 weeks
17. History of ketoacidosis
18. history of repeated urogenital infection
19. hemoglobinopathies, haemolytic anaemia, or chronic anaemia (haemoglobin concentration <12.0 g/dL)
20. presence of psychiatric disorder or new intake of antidepressant or antipsychotic agents(start within last 3 months)
21. Positive Screening for a severe depression (BDI ≥29)
22. history of hypersensitivity to the study drug or its ingredients
23. more than 5% weight loss in the last 3 months
24. Pregnant or breastfeeding women
25. Subject (male, female or intersexual) is not willing to use highly effective contraceptive methods during treatment and for 14 days (male or female) after the end of treatment (highly effective methods are defined as: combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner, sexual abstinence).

    Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the trial participant and that the vasectomized partner has received medical assessment of the surgical success.
26. Current participation in other interventional clinical trials or treatment with other IMPs within five times the half-life of the drug
27. Previous therapy with dapagliflozin or other drugs that can potentially lead to overlapping toxicities within five times the half-life of the drug
28. Patients who do not want to be informed about accidental findings
29. Any other clinical condition that would jeopardize subjects' safety or well-being while participating in this clinical trial
30. Patients will not be included in the study if, in the opinion of the investigator, participation leads to an unacceptable risk to their safety and well-being

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of remission of hyperglycemia | 6 months
  Frequency of individuals with prediabetes remission (normalization of fasting and 2h glucose concentrations) with dapagliflozin in comparison to treatment with placebo.

SECONDARY OUTCOMES:
Reduction of urinary albumine-creatinine ratio. | 1 month throuhg 6 months
  To test differences between the two treatment arms for reduction of urinary albumine-creatinine ratio.
Change in estimated glomerular filtration rate (eGFR) | 7 months
  To test differences between the two treatment arms for reduction in estimated glomerular filtration rate (eGFR).
Slopes over time of estimated glomerular filtration rate (eGFR). | baseline to 4 weeks, baseline to 7 months, 3 months to 7 months, baseline to 12 months
  To test differences between the two treatment arms for slopes over time of estimated glomerular filtration rate (eGFR).
Numbers of patients showing resolution of chronic kidney disease (CKD) | 3 months through 12 months
  To test differences between the two treatment arms for resolution of chronic kidney disease (CKD) for at least 3 months continuously: Urine Albumin Creatinin Ratio (uACR) < 30mg/g
Prediabetes remission maintenance | 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on remission of prediabetes as defined in the oGTT a fasting glucose <100 mg/dl and 2 h glucose <140 mg/dl at follow up

OTHER OUTCOMES:
Insulin sensitivity | 6 months, 12 months
  Baseline-adjusted insulin sensitivity at EoT using Insulin sensitivity: ISI-Matsuda/Oral glucose insulin sensitivity index.
Insulin secretion | 6 months, 12 months
  Baseline-adjusted insulin secretion at EoT using an estimate for insulin secretion: C-peptide0-30AUC/glucose0-30AUC.
Number of patients progressing to Type 2 Diabetes | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on the progression to T2DM as defined as a HbA1c ≥ 6.5
Change in body weight | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on change in body weight.
Change in BMI | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on BMI.
Change in whole body fat | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on whole body fat measures by magnetic resonance imaging.
Change in visceral fat | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on visceral fat measures by magnetic resonance imaging.
Change in liver fat | 6 months, 12 months
  Effects of 6 months reatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on liver fat measures by magnetic resonance spectroscopy.
Change in subcutaneous fat | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on subcutaneous fat measures by magnetic resonance imaging.
Arterial blood pressure | 6 months, 7 months, 12 months
  Baseline-adjusted arterial blood pressure at EoT
New onset or progress of neuropathy | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on new onset or progress of and neuropathy assessed by using the Rydel-Seiffer tuning fork and a 10 g monofilament
Quality of life using the Short Form Health Survey (SF)-36 questionnaire | 6 months, 12 months
  Effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on quality of life using the SF-36 questionnaire (scored on a 0 to 100 range; the higher the score, the higher quality of life)
Interaction between diabetes risk cluster and intervention for numbers of patients showing a resolution of Prediabetes | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on remission of prediabetes as defined a fasting glucose <100 mg/dl and 2 h glucose <140 mg/dl in the OGTT.
Interaction between diabetes risk cluster and intervention for change in albuminuria | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for kidney damage as shown by albuminuria in patients with CKD stage G1A2/G2A2 and prediabetes can be improved by a treatment with the SGLT2 inhibitor dapagliflozin (10mg/day) and lifestyle counselling compared to placebo and lifestyle counselling for 6 months calculated as mean of baseline-adjusted uACR measurements with dapagliflozin in comparison to treatment with placebo.
Interaction between diabetes risk cluster and intervention for change in estimated glomerular filtration rate (eGFR). | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention on estimated glomerular filtration rate (eGFR).
Interaction between diabetes risk cluster and intervention for slopes over time of estimated glomerular filtration rate (eGFR). | 4 weeks, 3 months, 6 months, 7 months, 12 months
  To test interaction between diabetes risk clusters and intervention on slopes over time of estimated glomerular filtration rate (eGFR).
Interaction between diabetes risk cluster and intervention for numbers of patients showing resolution of chronic kidney disease (CKD) | 3 months, 6 months, 7 months, 12 months
  To test interaction between diabetes risk clusters and intervention for resolution of chronic kidney disease (CKD) for at least 3 months continuously: Urine Albumin Creatinin Ratio (uACR) < 30mg/g
Interaction between diabetes risk cluster and intervention for insulin sensitivity. | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for baseline-adjusted insulin sensitivity at EoT using Insulin sensitivity: ISI-Matsuda/Oral glucose insulin sensitivity index.
Interaction between diabetes risk cluster and intervention for insulin secretion | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for baseline-adjusted insulin secretion at EoT using insulin secretion:C-peptide0-30AUC/glucose0-30AUC.
Interaction between diabetes risk cluster and intervention for number of patients progressing to Type 2 Diabetes | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on the progression to T2DM as defined as a HbA1c ≥ 6.5
Interaction between diabetes risk cluster and intervention for change in body weight | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on change in body weight.
Interaction between diabetes risk cluster and intervention for change in BMI. | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on BMI.
Interaction between diabetes risk cluster and intervention for change in whole body fat | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on whole body fat measures by magnetic resonance imaging.
Interaction between diabetes risk cluster and intervention for change in visceral fat | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on visceral fat measures by magnetic resonance imaging.
Interaction between diabetes risk cluster and intervention for change in liver fat | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on liver fat measures by magnetic resonance spectroscopy.
Interaction between diabetes risk cluster and intervention for change in subcutaneous fat | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on subcutaneous fat measures by magnetic resonance imaging.
Interaction between diabetes risk cluster and intervention for change in arterial blood pressure | 6 months, 7 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on the arterial blood pressure
Interaction between diabetes risk cluster and intervention on the new onset or progress of neuropathy | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on the new onset or progress of neuropathy assessed by using the Rydel-Seiffer tuning fork and a 10 g monofilament.
Interaction between diabetes risk cluster and intervention for change in quality of life | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on the quality of life using the SF-36 questionnaire (scored on a 0 to 100 range; the higher the score, the higher quality of life).
Small vessel density | 6 months, 12 months
  Change in small vessel density and junction-to-endpoint branches between baseline and EoT in the dapagliflozin versus placebo group as assessed by optoacustic imagingMyocardial function
Interaction between diabetes risk cluster and intervention on small vessel density | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for change in small vessel density and junction-to-endpoint branches between baseline and EoT in the dapagliflozin versus placebo group as assessed by optoacustic imagingMyocardial function
New onset or progress of diabetic retinopathy | 6 months, 12 months
  New onset or progress of retinopathy between baseline and EoT in the dapagliflozin versus placebo group. This will be assessed by a grading algorithm using the iCare DRSplus camera. Since macula edema at early stages cannot adequately be assessed with fundus pictures, we will assess maculopathies using optical coherence tomography
Interaction between diabetes risk cluster and intervention on the new onset or progress of diabetic retinopathy | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on the new onset or progress of retinopathy between baseline and EoT in the dapagliflozin versus placebo group. This will be assessed by a grading algorithm using the iCare DRSplus camera. Since macula edema at early stages cannot adequately be assessed with fundus pictures, we will assess maculopathies using optical coherence tomography.
Composition of the gut microbiome | 3 months, 6 months, 7 months, 12 months
  Change in gut microbial community and gene abundances within and between intervention and placebo groups over time using next generation sequencing data and machine learning algorithms
Interaction between diabetes risk cluster and intervention for composition of the gut microbiome | 3 months, 6 months, 7 months, 12 months
  To test interaction between diabetes risk clusters and intervention change in gut microbial community and gene abundances within and between intervention and placebo groups over time using next generation sequencing data and machine learning algorithms
Urinary metabolite signature of SGLT2 inhibitors | 6 months, 12 months
  Changes in urinary metabolites within and between intervention and placebo groups over time using MS-based metabolomics and machine learning algorithms
Interaction between diabetes risk cluster and intervention for urinary metabolite signature of SGLT2 inhibitors | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention changes in urinary metabolites within and between intervention and placebo groups over time using MS-based metabolomics and machine learning algorithms
Myocardial function shown by left ventricular mass index | 6 months, 12 months
  Effects of dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on left ventricular mass index assessed via cardiac magnetic resonance imaging
Interaction between diabetes risk cluster and intervention on Myocardial function shown by left ventricular mass index | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on left ventricular mass index assessed via cardiac magnetic resonance imaging.
Myocardial function shown by systolic myocardial function | 6 months, 12 months
  Effects of dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on systolic myocardial function assessed via cardiac magnetic resonance imaging.
Interaction between diabetes risk cluster and intervention on Myocardial function shown by systolic myocardial function | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on systolic myocardial function assessed via cardiac magnetic resonance imaging.
Myocardial function shown by diastolic myocardial function | 6 months, 12 months
  Effects of dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on diastolic myocardial function assessed via cardiac magnetic resonance imaging.
Interaction between diabetes risk cluster and intervention on Myocardial function shown by diastolic myocardial function | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on diastolic myocardial function assessed via cardiac magnetic resonance imaging.
Health economic evaluation shown by incremental cost-effectiveness ratio | 6 months, 12 months
  Conducting a health economic evaluation from the perspective of the statutory health insurance and society in from of a cost-effectiveness analysis
Interaction between diabetes risk cluster and intervention on health economic evaluation shown by incremental cost-effectiveness ratio | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on health economic evaluation shown by incremental cost-effectiveness ratio of a cost-effectiveness analysis
Health economic evaluation shown by incremental cost-utility ratio | 6 months, 12 months
  Conducting a health economic evaluation from the perspective of the statutory health insurance and society in from of a cost-utility analysis
Interaction between diabetes risk cluster and intervention on health economic evaluation shown by incremental cost-utility ratio | 6 months, 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on health economic evaluation shown by incremental cost-utility ratio of a cost-utility analysis
Changes in risk preferences | 6 months, 12 months
  To test differences between the two treatment arms for the risk preferences
Changes in time preferences | 6 months, 12 months
  To test differences between the two treatment arms for the time preferences
Interaction between diabetes risk cluster and intervention on prediabetes remission maintenance | 12 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on remission of prediabetes as defined in the oGTT a fasting glucose <100 mg/dl and 2 h glucose <140 mg/dl at follow up.
Interaction between diabetes risk cluster and intervention on the risk preferences | 6 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on change of risk preferences
Interaction between diabetes risk cluster and intervention on the risk preferences | 6 months
  To test interaction between diabetes risk clusters and intervention for effects of 6 months treatment with dapagliflozin 10 mg and lifestyle counseling compared to placebo and lifestyle intervention on change of time preferences

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (9):
  - Charité Universitätsmedizin Berlin, Klinik für Endokrinologie und Stoffwechselmedizin, Berlin
  - Universitätsstudienzentrum für Stoffwechselerkrankungen , Medizinische Klinik und Poliklinik III, Dresden
  - German Diabetes Center, Leibniz-Center for Diabetes Research at the Heinrich-Heine-University Duesseldorf, Düsseldorf
  - Heidelberg University Hospital - Department of Endocrinology and Metabolism, Heidelberg
  - Medizinische Klinik und Poliklinik III - Bereich Endokrinologie, Leipzig
  - Medizinische Klinik I, UKSH Campus LübeckAG Meyhöfer - Endocrinology, Diabetes & Metabolism, Lübeck
  - Diabetes Center Med. Klinik und Poliklinik IV, Klinikum der Universität München, LMU, München
  - Institut für Ernährungsmedizin, Technische Universität München, München
  - University Hospital Tuebingen, Otfried-Mueller Str. 10, Tübingen